CLINICAL TRIAL: NCT00819741
Title: A 16-week, Open-label, Multicentre, Randomised, Parallel Study to Evaluate Efficacy and Safety of Repaglinide and Metformin Combination Therapy Compared to Repaglinide Monotherapy in Chinese OAD Naive Type 2 Diabetic Patients
Brief Title: Comparison of the Blood Sugar Lowering Effect Between Repaglinide Plus Metformin and Repaglinide Alone in Type 2 Diabetics Not Previously Treated With Oral Sugar-lowering Drugs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGEE-3705
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Results first posted 2010-12-08 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Repaglinide + metformin (Experimental): Initial dose of repaglinide 1mg plus metformin 500mg once daily. During the dose titration period of 6 weeks, the dose could be titrated up to repaglinide 4 mg and metformin 500 mg three times daily, according to fasting glucose values. The minimal dose was repaglinide 1 mg plus metformin 500 mg three times daily.
  Interventions: Drug: repaglinide; Drug: metformin
- Repaglinide (Active Comparator): Initial dose of repaglinide 1 mg three times daily. During the dose titration period of 6 weeks, the dose of repaglinide could be titrated up to 4 mg three times daily, according to fasting glucose values. The minimal dose was repaglinide 1 mg three times daily.
  Interventions: Drug: repaglinide

INTERVENTIONS:
Drug: repaglinide — The dose was started from repaglinide 1 mg plus metformin 500 mg once daily. During the dose titration period, the dose could be titrated up to repaglinide 4 mg and metformin 500mg three times daily, according to fasting glucose. the minimal dose was repaglinide 1 mg plus metformin 500 mg three times daily
  Arms: Repaglinide + metformin
Drug: metformin — The dose was started from repaglinide 1 mg plus metformin 500 mg once daily. During the dose titration period, the dose could be titrated up to repaglinide 4 mg and metformin 500 mg three times daily, according to fasting glucose. the minimal dose was repaglinide 1 mg plus metformin 500 mg three times daily
  Arms: Repaglinide + metformin
Drug: repaglinide — The dose was started from repaglinide 1 mg three times daily. During the dose titration period, the dose of repaglinide could be titrated up to 4 mg three times daily, according to fasting glucose.
  Arms: Repaglinide

SUMMARY:
This trial is conducted in Asia. The aim of this clinical trial is to investigate the blood sugar lowering effect of repaglinide plus metformin as initial treatment compared to repaglinide alone in Chinese subjects with type 2 diabetes having an HbA1c (glycosylated haemoglobin A1c) over 8.5 % and who never have taken oral sugar-lowering drugs before. The associated unfavourable events including low blood sugar episodes between the two treatments are also compared.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* Never taken oral antidiabetic drugs before
* HbA1c greater than 8.5 %
* BMI (Body Mass Index) less than or equal to 35 kg/m^2

Exclusion Criteria:

* Known or suspected allergy to repaglinide, metformin, or any of the excipients in the medications
* Taken an investigational drug in another clinical trial within 4 weeks prior to this trial
* Impaired liver function, defined as ASAT (aspartate aminotransferase) or ALAT (alanine aminotransferase) equal to or greater than 2 times upper normal limit
* Have a clinically significant, active disease of the gastrointestinal, pulmonary, neurological, renal, genitourinary, and haematological systems
* Severe uncontrolled or untreated hypertension (sitting diastolic blood pressure (BP) equal to or greater than 100 mmHg or systolic BP equal to or greater than 180 mmHg)
* Impaired renal function
* Acute or chronic acidosis or if there are plans to have a radiographic material containing iodine
* Have a clinically significant, active cardiovascular disease, or decompensated heart failure
* Treatment with systemic corticosteroids within the past two months prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2009-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (11):
- China (11):
  - Novo Nordisk Investigational Site, Fuzhou, Fujian
  - Novo Nordisk Investigational Site, Nanjing, Jiangsu
  - Novo Nordisk Investigational Site, Suzhou, Jiangsu
  - Novo Nordisk Investigational Site, Wuxi, Jiangsu
  - Novo Nordisk Investigational Site, Nanchang, Jiangxi
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality
  - Novo Nordisk Investigational Site, Hangzhou, Zhejiang
  - Novo Nordisk Investigational Site, Wenzhou, Zhejiang
  - Novo Nordisk Investigational Site, Hangzhou
  - Novo Nordisk Investigational Site, Nantong
  - Novo Nordisk Investigational Site, Shanghai

REFERENCES:
- [Result] Wang W, Bu R, Su Q, Liu J, Ning G. Randomized study of repaglinide alone and in combination with metformin in Chinese subjects with type 2 diabetes naive to oral antidiabetes therapy. Expert Opin Pharmacother. 2011 Dec;12(18):2791-9. doi: 10.1517/14656566.2011.602341. Epub 2011 Jul 22. PMID 21780853
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 17 sites in China.
Pre-assignment Details: Between screening and treatment with trial drug, subjects were assessed for eligibility and were randomised to one of two treatment arms. After start of treatment, all the subjects underwent a 6-week dose titration period followed by a 10-week maintenance period. A subgroup of 50 subjects from each treatment group was chosen.
Period: Overall Study
Arm/Group | Repaglinide + Metformin | Repaglinide
Started | 218 | 215
Exposed to Drug | 218 | 214 (One subject after randomisation was not exposed to the treatment due to non-compliance)
Completed | 196 | 201
Not Completed | 22 | 14
Not completed — Adverse Event | 5 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Protocol Violation | 3 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Unclassified | 6 | 0
Not completed — Reasons unknown | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Repaglinide + Metformin | Repaglinide | Total
Number analyzed (Participants) | 218 | 214 | 432
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (9.6) | 49.4 (10.0) | 49.9 (10.0)
Gender [Count of Participants; unit: Participants]
  Female | 60 | 59 | 119
  Male | 158 | 155 | 313
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 218 | 214 | 432
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] — BMI (Body Mass Index)
  kg/m^2 | 24.50 (2.97) | 24.44 (3.05) | 24.47 (3.00)
Weight [Mean (Standard Deviation); unit: kg] | 68.3 (10.8) | 68.2 (11.0) | 68.3 (10.9)
Duration of diabetes [Mean (Standard Deviation); unit: months] — Number of months since dignosis
  months | 0.14 (0.73) | 0.28 (1.57) | 0.21 (1.22)
HbA1c [Mean (Standard Deviation); unit: percentage (%) of total haemoglobin] — Glycosylated haemoglobin A1c
  percentage (%) of total haemoglobin | 10.91 (1.45) | 10.73 (1.50) | 10.82 (1.48)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin A1c (HbA1c)
Description: Calculated as an estimate of the mean change in HbA1c after 16 weeks of treatment.
Time Frame: week -2 (screening), week 16
Population: Intention-to-Treat analysis set (ITT) is all subjects who entered the trial treatment period and exposed to at least one dose of trial product.
Measure: Least Squares Mean (Standard Error); unit: percentage (%) of total haemoglobin
Arm/Group | Repaglinide + Metformin | Repaglinide
Number analyzed (Participants) | 212 | 209
percentage (%) of total haemoglobin | -4.450 (0.070) | -4.148 (0.071)
Statistical Analysis 1: Comparison: Repaglinide + Metformin vs Repaglinide; The non-inferiority margin for HbA1c was set to 0.4%. The null hypothesis (H0) was: H0: HbA1c of repaglinide + metformin therapy after 16 weeks of treatment - HbA1c of repaglinide monotherapy after 16 weeks of treatment ≥0.4% Against the alternative hypothesis (H1): H1: HbA1c of repaglinide + metformin therapy after 16 weeks of treatment - HbA1c of repaglinide monotherapy after 16 weeks of treatment <0.4%; Test type: Non-Inferiority or Equivalence — If non-inferiority was shown (that was if H0 was rejected), then superiority of repaglinide and metformin combination therapy compared to repaglinide monotherapy would be claimed if the upper limit of the 95% CI for the difference was lower than 0%. The non-inferiority margin for HbA1c was set to 0.4%; ANCOVA; Estimated treatment difference, LS Mean = -0.302, 95% CI [-0.491 to -0.114], Standard Error of Mean 0.0096

2. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Calculated as an estimate of the mean change in fasting plasma glucose after 16 weeks of treatment.
Time Frame: week 0, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Repaglinide + Metformin | Repaglinide
Number analyzed (Participants) | 211 | 209
mmol/L | -4.646 (0.129) | -3.982 (0.130)

3. Secondary Outcome: Change in 2-hour Postprandial Plasma Glucose
Description: Calculated as an estimate of the mean change in 2-hour postprandial plasma glucose following a standard test meal after 16 weeks of treatment
Time Frame: Week 0, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Repaglinide + Metformin | Repaglinide
Number analyzed (Participants) | 210 | 204
mmol/L | -7.525 (0.237) | -6.794 (0.242)

4. Secondary Outcome: Change in 7-point Plasma Glucose Profile
Description: Calculated as an estimate of the mean change in 7-point (before breakfast, 2 hours after breakfast, before lunch, 2 hours after lunch, before dinner, 2 hours after dinner, bedtime) plasma glucose profile after 16 weeks of treatment.
Time Frame: Week 0, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Repaglinide + Metformin | Repaglinide
Number analyzed (Participants) | 218 | 214
mmol/L
  Before breakfast, N=204, 199 | -4.99 (0.11) | -4.58 (0.12)
  2 hours after breakfast, N=206, 201 | -7.85 (0.23) | -7.40 (0.24)
  Before lunch, N=203, 200 | -6.85 (0.18) | -6.28 (0.18)
  2 hours after lunch, N=204, 201 | -8.00 (0.21) | -6.98 (0.21)
  Before dinner N=204, 202 | -5.62 (0.17) | -5.09 (0.17)
  2 hours after dinner N=204, 199 | -7.13 (0.21) | -5.70 (0.22)
  Bedtime N=195, 188 | -6.93 (0.19) | -5.82 (0.19)
  Average N=207, 202 | -6.78 (0.14) | -5.99 (0.14)

5. Secondary Outcome: Change in Fasting Serum Insulin
Description: Calculated as an estimate of the mean change in fasting serum insulin after 16 weeks of treatment.
Time Frame: Week 0, week 16
Population: Intention-to-Treat analysis set (ITT) is all subjects who entered the trial treatment period and exposed to at least one dose of trial product. A total of 100 subjects (50 per study group) out of the total subjects were randomly selected in the trial. Four trial sites were selected for the subgroup study.
Measure: Least Squares Mean (Standard Error); unit: mU/L
Arm/Group | Repaglinide + Metformin | Repaglinide
Number analyzed (Participants) | 49 | 46
mU/L | 3.163 (1.801) | 5.694 (1.872)

6. Secondary Outcome: Change in 2-hour Postprandial Serum Insulin
Description: Calculated as an estimate of the mean change in 2-hour postprandial serum insulin after 16 weeks of treatment.
Time Frame: Week 0, week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mU/L
Arm/Group | Repaglinide + Metformin | Repaglinide
Number analyzed (Participants) | 49 | 44
mU/L | 34.083 (6.731) | 28.548 (7.132)

7. Secondary Outcome: Change in Fasting Serum C-peptide
Description: Calculated as an estimate of the mean change in fasting serum C-peptide after 16 weeks of treatment
Time Frame: Week 0, week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: ng/ml
Arm/Group | Repaglinide + Metformin | Repaglinide
Number analyzed (Participants) | 49 | 46
ng/ml | 0.041 (0.123) | 0.405 (0.128)

8. Secondary Outcome: Change in 2-hour Postprandial Serum C-peptide
Description: Calculated as an estimate of the mean change in 2-hour postprandial serum C-peptide after 16 weeks of treatment
Time Frame: Week 0, week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: ng/ml
Arm/Group | Repaglinide + Metformin | Repaglinide
Number analyzed (Participants) | 49 | 44
ng/ml | 2.301 (0.347) | 2.081 (0.369)

9. Secondary Outcome: Hypoglycaemic Episodes
Description: Number of hypoglycaemic episodes from Week 0 to Week 16, defined as major, minor or symptoms only. Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose below 3.1 mmol/L. Symptoms only if able to treat her/himself and no plasma glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L.
Time Frame: Weeks 0-16
Population: Safety analysis set was defined as all randomised and exposed subjects.
Measure: Number; unit: episodes
Arm/Group | Repaglinide + Metformin | Repaglinide
Number analyzed (Participants) | 218 | 214
episodes
  Major | 0 | 0
  Minor | 41 | 16
  Symptoms only | 90 | 71

10. Secondary Outcome: Change in Blood Pressure
Description: Calculated as the mean change in diastolic and systolic blood pressure after 16 weeks of treatment
Time Frame: Week 0, week 16
Population: Safety analysis set was defined as all randomised and exposed subjects.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Repaglinide + Metformin | Repaglinide
Number analyzed (Participants) | 196 | 201
mmHg
  Blood pressure diastolic | -1.0 (8.8) | -0.9 (9.5)
  Blood pressure systolic | -1.5 (14.3) | -1.4 (14.2)

11. Secondary Outcome: Physical Examinations
Description: The number of subjects having a physical examination event that changed from 'Normal' or 'Abnormal, not clinically significant' to 'Abnormal, clinically significant'. Physical examination included cardiovascular system, respiratory system, musculoskeletal system, nervous system and abdomen.
Time Frame: Week -2, week 16
Population: Safety analysis set was defined as all randomised and exposed subjects.
Measure: Number; unit: Subjects
Arm/Group | Repaglinide + Metformin | Repaglinide
Number analyzed (Participants) | 218 | 214
Subjects | 3 | 0

12. Secondary Outcome: ECG (ElectroCardioGram)
Description: The number of subjects having a electrocardiogram (ECG) that changed from 'Normal' or 'Abnormal, not clinically significant' to 'Abnormal, clinically significant'. 'Abnormal, Clinically significant' is an abnormality that suggests a disease and/or organ toxicity and is of a severity, which requires active management.
Time Frame: Week -2, week 16
Population: Safety analysis set was defined as all randomised and exposed subjects.
Measure: Number; unit: Subjects
Arm/Group | Repaglinide + Metformin | Repaglinide
Number analyzed (Participants) | 218 | 214
Subjects | 3 | 2

13. Secondary Outcome: Biochemistry: Alanine Aminotransferase (ALAT)
Description: The number of subjects having a change in Alanine Aminotransferase (ALAT) from 'Normal' or 'Abnormal, not clinically significant' to 'Abnormal, clinically significant'. 'Abnormal, Clinically significant' is an abnormality that suggests a disease and/or organ toxicity and is of a severity, which requires active management.
Time Frame: Week -2, week 16
Population: Safety analysis set was defined as all randomised and exposed subjects.
Measure: Number; unit: Subjects
Arm/Group | Repaglinide + Metformin | Repaglinide
Number analyzed (Participants) | 218 | 214
Subjects | 4 | 5

14. Secondary Outcome: Biochemistry: Alanine Aminotransferase (ASAT)
Description: The number of subjects having a change in Aspartate Aminotransferase (ASAT) from 'Normal' or 'Abnormal, not clinically significant' to 'Abnormal, clinically significant'. 'Abnormal, Clinically significant' is an abnormality that suggests a disease and/or organ toxicity and is of a severity, which requires active management.
Time Frame: Week -2, week 16
Population: Safety analysis set was defined as all randomised and exposed subjects.
Measure: Number; unit: Subjects
Arm/Group | Repaglinide + Metformin | Repaglinide
Number analyzed (Participants) | 218 | 214
Subjects | 2 | 4

15. Secondary Outcome: Haematology: Haemoglobin
Description: Haemoglobin was measured. The number of subjects having a change in Haemoglobin measurement from 'Normal' or 'Abnormal, not clinically significant' to 'Abnormal, clinically significant' 'Abnormal, Clinically significant' is an abnormality that suggests a disease and/or organ toxicity and is of a severity, which requires active management.
Time Frame: Week -2, week 16
Population: Safety analysis set was defined as all randomised and exposed subjects.
Measure: Number; unit: Subjects
Arm/Group | Repaglinide + Metformin | Repaglinide
Number analyzed (Participants) | 218 | 214
Subjects | 1 | 0

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time span of 16 weeks.
Description: The safety analysis set contains all randomised subjects exposed to at least one dose of trial drug(s).
Arm/Group | Repaglinide + Metformin | Repaglinide
Serious Adverse Events (participants affected / at risk) | 0/218 | 1/214
Other Adverse Events (participants affected / at risk) | 0/218 | 0/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Repaglinide + Metformin (N=218) | Repaglinide (N=214)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right to not release data until specified milestones, e.g. when the clinical trial report is available. At the end of the trial, one or more manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property.